CLINICAL TRIAL: NCT07297030
Title: A Prospective Single-Arm Phase II Clinical Study of Neoadjuvant Short-Course Radiotherapy With Simultaneous Integrated Boost Combined With Capecitabine-Oxaliplatin and PD-1 Inhibitor Therapy in High-Risk Locally Advanced Rectal Cancer
Brief Title: SIB-RT Combined With CAPOX and PD-1 for High-Risk Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, M.D., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-38
Record Dates: First submitted 2025-07-13; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer
Keywords: SIB; PD-1; neoadjuvant chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIB-SCRT+CAPOX+PD-1 (Experimental): Patients received neoadjuvant treatment consisting of SIB-SCRT ( PTV-GTV 31Gy/5F/6.2Gy) followed by sintilimab (3mg/kg intravenous drip on day 1; every 3-week cycle for two cycles) combined with CAPOX (oxaliplatin 130 mg/m2 intravenous infusion over 2 h on day 1, capecitabine 1000 mg/m2 orally twice daily from day 1-14, in every 3-week cycle for two cycles) 1 week later.
  Interventions: Radiation: SIB-SCRT; Drug: CAPOX; Drug: Immunotherapy

INTERVENTIONS:
Radiation: SIB-SCRT — The pelvic lymphatic drainage regions receive 25 Gy in 5 fractions (5 Gy per fraction). A ssequential boost to a total dose of 30 Gy in 6 fractions is delivered to the primary tumour and any radiologically suspicious lymph nodes.
Drug: CAPOX — * Oxaliplatin 130 mg/m² intravenously on day 1.
  * Capecitabine 1,000 mg/m² orally twice daily on days 1-14.
Drug: Immunotherapy — - Tislelizumab 200 mg intravenously on day 1.

SUMMARY:
The biological effective dose of short-course radiotherapy is relatively lower compared to long-course radiotherapy, which may lead to an increased local recurrence rate in patients with mid to low rectal cancer who are at high risk of locally advanced disease due to insufficient radiation dose. Combining short-course radiotherapy with simultaneous integrated boost (SIB) and immunotherapy-chemo regimens could potentially further enhance tumor regression and improve local control, providing a promising treatment option for high-risk locally advanced rectal cancer patients. Therefore, this clinical trial aims to explore the safety and effectiveness of a short-course SIB radiotherapy regimen combined with immunotherapy and chemotherapy as neoadjuvant treatment for locally advanced rectal cancer, based on short-course radiotherapy combined with chemotherapy and immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must voluntarily agree to join this study and sign an informed consent form.
* Age at the time of signing the informed consent form must be between 18 and 75 years.
* Histologically confirmed diagnosis of rectal adenocarcinoma.
* High-risk locally advanced pMMR/MSS rectal cancer, categorized according to the AJCC/UICC 8th edition clinical staging and in reference to the inclusion criteria of the RAPIDO study, must meet at least one of the following conditions: cT4 stage, cN2 stage, involvement of the mesorectal fascia (MRF), or presence of laterally enlarged lymph nodes, with M0 status.
* The inferior margin of the tumor must be ≤10 cm from the anal verge.
* No prior anti-cancer treatment for rectal cancer (including local-regional and systemic therapy).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1.
* At least one measurable lesion according to RECIST v1.1 criteria.
* Normal function of major organs without severe abnormalities in hematological, cardiovascular, pulmonary, hepatic, renal, or bone marrow function; laboratory tests must meet the following requirements:

Hemoglobin (Hb) ≥ 70 g/L; White blood cell count (WBC) ≥ 3.0 × 10^9/L; Neutrophil count (NEUT) ≥ 1.5 × 10^9/L; Platelet count (PLT) ≥ 100 × 10^9/L; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times the upper limit of normal (ULN); Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Renal function (serum creatinine, sCr) level ≤ 1.5 times the upper limit of normal (ULN).

Exclusion Criteria:

* Evidence of distant metastasis.
* Recurrent rectal cancer.
* Documented allergy to the investigational drug and/or its excipients.
* Contraindications to radiotherapy and/or chemotherapy.
* Women who are pregnant or breastfeeding.
* A history of other malignancies.
* Patients who have participated in other clinical trials involving investigational drugs within the last 6 months.
* Patients deemed inappropriate for inclusion in this study as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
The Complete Response (CR) rate | 3 months
  The Complete Response (CR) rate refers to the sum of the pathological Complete Response (pCR) rate, defined as the absence of residual cancer cells in the surgical resection specimen observed microscopically, and the probability of patients achieving clinical Complete Response (cCR) who then undergo a watchful waiting (W&W) approach. The primary endpoint of my study is the CR rate.

SECONDARY OUTCOMES:
Rate of ≥Grade 3 toxicities | 3 months
  This endpoint measures the incidence of adverse events classified as Grade 3 or higher according to the Common Terminology Criteria for Adverse Events (CTCAE). A Grade 3 toxicity indicates a severe reaction that significantly affects the patient's daily activities and typically requires medical intervention. Monitoring the rate of these serious toxicities will help evaluate the safety profile of the treatment regimen, including neoadjuvant short-course radiotherapy combined with simultaneous integrated boost, immunotherapy, and chemotherapy, in patients with high-risk locally advanced rectal cancer. Assessing these toxicities is critical for understanding the balance between therapeutic efficacy and tolerability in this patient population.
3-Year Disease-Free Survival Rate (3yDFS%) | 3 years
  The 3-Year Disease-Free Survival Rate (3yDFS%) refers to the percentage of patients who do not experience any disease progression within three years after completing the treatment.
3-Year Locoregional Recurrence-Free Survival Rate (3yLRFS%) | 3 years
  The 3-Year Locoregional Recurrence-Free Survival Rate (3yLRFS%) is defined as the percentage of patients who remain free from locoregional recurrence of cancer for three years after completing the treatment.
3-Year Overall Survival Rate (3yOS%) | 3 years
  This endpoint refers to the percentage of patients who are still alive three years after receiving the treatment, regardless of disease status.
Surgical Complications | 6 months
  This endpoint assesses the occurrence of adverse events related to the surgical procedure performed on patients with high-risk locally advanced rectal cancer. Surgical complications may include infections, bleeding, anastomotic leaks, and any other significant morbidity that may influence the patient's postoperative recovery.
Quality of Life (QoL) | 3 years
  This endpoint evaluates the overall well-being of patients following treatment, focusing on their physical, emotional, and social health. Quality of Life assessments will be performed using validated questionnaires, such as the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). This scale comprises multiple dimensions, including physical functioning, emotional functioning, and social functioning, with scores ranging from 0 to 100, where higher scores indicate better quality of life.
  The assessments will provide insights into patients' functional status and any changes in health-related quality of life resulting from the treatment regimen. Understanding QoL outcomes is essential for assessing the patient-centered effectiveness of the therapeutic approach and ensuring that treatment strategies not only target disease control but also support the overall well-being of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No